CLINICAL TRIAL: NCT03814837
Title: A Study for the Ocular Toxocariasis in the Patients Who Were Diagnosed With the Pulmonary Toxocariasis, and Ocular Toxocariasis Cohort: TOXOCARA Study
Brief Title: A Study for the Ocular Toxocariasis Patients With the Pulmonary Toxocariasis, and Ocular Toxocariasis Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ulsan (Other)
Collaborators: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Kwang Won Seo, Associate professor, division of pulmonology, dept. of internal medicine, University of Ulsan
Other Study IDs: UUH 2017-06-012-001
Record Dates: First submitted 2019-01-09; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Toxocariasis; Ocular Toxocariasis; Pulmonary Toxocariasis; Ground Glass Opacity (GGO); Toxocara Canis Infection (Canine Roundworms); Law Liver; Law Meat; Serum Toxocara Antibody; Toxocara Larva Migrans
MeSH Terms: conditions — Toxocariasis; Larva Migrans; Toxocara canis infection (canine roundworms)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TOXOCARA Study is a prospective observational cohort study. The aim of this study is to evaluate the incidence of ocular toxocariasis (OT) associated with pulmonary toxocariasis (PT) in patients with chest diagnostic image tests (chest X-ray, chest CT) with migrating ground glass opacity or nodular lesions. Also a cohort study is to track the results of treatment for diagnosed ocular toxocariasis (OT) patients.

DETAILED DESCRIPTION:
Toxocara canis (also known as dog roundworm) is wide-reaching parasite of dogs and other canids. It can spread between animals such as cats, pigs and cows by ingestion of worm eggs from the feces of an infected animal.

In humans, two pathways of infection are known: first, ingestion of the eggs and second, larvae encapsulated in the tissues of the infected animal.

The encapsulated larvae hatch in the small intestine and pass through the barrier to the portal vein, the liver, the lung, the eye, etc. and remain as encapsulated larvae or survive for a period of time.

Infection into humans has been reported through ingestion of uncooked liver of cows, pigs, sheep, chickens, and meat (muscle).

When encapsulated larvae migrate to the body such as lungs, eosinophils activate and proliferate to eliminate the parasites.

They can be expressed as ground glass opacity (GGO) or nodular lesion by aggregated eosinophils, which are mistaken for lung cancer or pneumonia to be investigated.

Asthma exacerbation, cough and other symptoms of respiratory system could be revealed, but often asymptomatic.

In this study, the investigators defined pulmonary toxocariasis (PT) as a positive form of serum toxocara Ab and migrating pulmonary GGOs or nodular lesions in chest diagnostic image tests (chest X-ray, chest CT) from the patient.

Also ocular toxocariasis (OT) is defined by the clinical manifestation of intraocular infection by Toxocara larvae with a positive result of serum toxocara Ab.

Clinical manifestations of OT may also cause blindness of peripheral granuloma, optic neuritis, chorioretinitis, conjunctivitis, keratitis, iridocyclitis and cataract.

The investigators want to investigate the incidence of OT associated with PT in patients with chest diagnostic image tests (chest X-ray, chest CT) with migrating GGOs or nodular lesions. Also a cohort study is to track the results of treatment for diagnosed OT patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Patient who has positive result of Toxocara Ab
* Patient who has history of eating of law animal liver or meat
* Patient who has the chest diagnostic image tests (chest X-ray, chest CT) with migrating ground glass opacity or nodular lesions.

Exclusion Criteria:

* Age < 18 years
* Pregnant woman
* Malignant patient
* Patient who has pulmonary infectious lesion such as pneumonia, fungus and tuberculosis
* Patients who were diagnosed by benign or malignant pulmonary nodule
* Patient who was not consented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators defined pulmonary toxocariasis (PT) as a positive form of serum toxocara Ab and migrating pulmonary GGOs or nodular lesions.
  Ocular toxocariasis (OT) is defined by the clinical manifestation of intraocular infection by Toxocara larvae and a positive form of serum toxocara Ab.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pulmonary toxocariasis (PT) | at baseline
  Patients who have a positive result of serum toxocara Ab and migrating pulmonary GGOs or nodular lesions and history of eating of law animal liver or meat or history of having the pets such as dogs and cats.
Number of patients with ocular toxocariasis (OT) | at baseline
  Patients who have the clinical manifestation of intraocular infection by Toxocara larvae and a positive result of serum toxocara Ab and history of eating of law animal liver or meat. (and/or migrating pulmonary GGOs or nodular lesions) or history of having the pets such as dogs and cats.
Number of patients with ocular toxocariasis (OT) among the patients with pulmonary toxocariasis (PT), | at baseline
  Patients who have ocular toxocariasis (OT) with pulmonary toxocariasis (PT)

SECONDARY OUTCOMES:
Incidence of Cysticercosis | at baseline
  Patient who have a positive result of serum cysticercosis Ab and history of eating of law animal liver or meat. (and/or migrating pulmonary GGOs or nodular lesions)
Incidence of Sparganosis | at baseline
  Patient who have a positive result of serum sparganum Ab and history of eating of law animal liver or meat. (and/or migrating pulmonary GGOs or nodular lesions)
Incidence of Clonorchiasis | at baseline
  Patient who have a positive result of serum clonorchis sinensis Ab and history of eating of the law freshwater fish or its cuisine. (and/or migrating pulmonary GGOs or nodular lesions)
Incidence of Paragonimiasis | at baseline
  Patient who have a positive result of serum paragonimus westermani Ab and history of eating of the law freshwater crabs or crayfish or its cuisine. (and/or migrating pulmonary GGOs or nodular lesions)
Incidence of Anisakiasis | at baseline
  Patient who have a positive result of serum anisakis Ab and history of eating of the law oceanic fish or its cuisine. (and/or migrating pulmonary GGOs or nodular lesions)
Clinical course of the patients with ocular toxocariasis (OT) after treatment | 3 years
  Follow-up : ocular toxocariasis cohort (clinical course of the patients with ocular toxocariasis (OT) after treatment by ophthalmologists)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Won Seo, M.D., Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, 877 Bangeojin Sunwhando-ro, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03814837/Prot_SAP_000.pdf